CLINICAL TRIAL: NCT00755118
Title: Phase II Study Of Weekly Administration Oxaliplatin Plus 5-Fu/Lv (Aio Regimen) Plus Bevacizumab, Alternative With Irinotecan Plus 5-Fu/Lv(Aio Regimen) Plus Cetuximab, As Salvage Treatment In Pretreated Patients With Mcrc
Brief Title: Lohp, 5-Fu/Lv and Bevacizumab, Alternative With Cpt-11, 5-Fu/Lv and Cetuximab In Metastatic Crc
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to poor Accrual
Sponsor: University Hospital of Crete (Other)
Responsible Party: Principal Investigator, Vassilis Georgoulias, MD, MD, University Hospital of Crete
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT/08.28
Record Dates: First submitted 2008-09-17; First posted 2008-09-18 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Colorectal Cancer
Keywords: Metastatic colorectal cancer; Second line; Irinotecan; Cetuximab; Bevacizumab
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Oxaliplatin; Fluorouracil; Leucovorin; Bevacizumab; Irinotecan; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): LoHP/AIO/Avastin->CPT-11/AIO/Erbitux
  Interventions: Drug: Oxaliplatin; Drug: 5-Fluorouracil; Drug: Leucovorin; Drug: Bevacizumab; Drug: Irinotecan; Drug: Cetuximab

INTERVENTIONS:
Drug: Oxaliplatin — Oxaliplatin (I.V) 85mg/m2 on week 1 and week 3 every six weeks for 2 continuously until disease progression or the appearance of unacceptable toxicity
  Other Names: Eloxatin; LoHP
Drug: 5-Fluorouracil — 5-Fluorouracil (I.V) 1750mg/m2 on week 1,2,3 and 4 every six weeks for 2 continuously until disease progression or the appearance of unacceptable toxicity
  Other Names: 5-FU
Drug: Leucovorin — Leucovorin (I.V) 500mg/m2 on week 1,2,3 and 4 every six weeks for 2 continuously until disease progression or the appearance of unacceptable toxicity
  Other Names: LV
Drug: Bevacizumab — Bevacizumab (I.V) 10mg/Kg on week 1 and week 3 every six weeks for 2 continuously until disease progression or the appearance of unacceptable toxicity
  Other Names: Avastin
Drug: Irinotecan — Irinotecan (I.V) 110mg/m2 on week 2 and week 4 every six weeks for 2 continuously until disease progression or the appearance of unacceptable toxicity
  Other Names: CPT-11; Campto
Drug: Cetuximab — Cetuximab (I.V) 500mg/m2 on week 2 and week 4 every six weeks for 2 continuously until disease progression or the appearance of unacceptable toxicity
  Other Names: Erbitux

SUMMARY:
The aim of this study is to evaluate the efficacy of the effective drugs in a alternating chemotherapy schedules in pretreated patients with mCRC, who have received all effective drugs.

DETAILED DESCRIPTION:
Colorectal cancer is a major cause of death worldwide and is ranked third in incidence and deaths from cancer in the USA for men and women. Incidence and mortality have been decreasing steadily in past decades, with 5-year survival for patients diagnosed in 1996-2002, being about 65%.

Although curative surgical resection is possible in 70-80% of patients at diagnosis, almost half of them will develop local or/and metastatic recurrence and will die of the disease.

There are currently three active cytotoxic agents that have been shown to be effective in the treatment of advanced colorectal cancer: 5-Fluorouracil combined with Leucovorin (5-FU/LV), Irinotecan and Oxaliplatin. During the last few years, the median overall survival of patients with advanced CRC has been substantially increased from 12 months to about 21-22 months, when combination of these chemotherapeutic agents are administered. Combinations of 5-Fluorouracil/Leucovorin (5-FU/LV) either as bolus (Roswell Park) or infusional administration (De Gramont schedule) r weekly infusional (AIO regimen), combined with Irinotecan or Oxaliplatin accepted as the mainstay of first line treatment.

The advent of targeted therapy further expanded treatment options for patients with mCRC.In particular, inhibition of Epidermal Growth Factor Receptor (EGFR) and angiogenesis by blocking Vascular Endothelial Growth Factor (VEGF) using monoclonal antibodies, led to further improvement in the outcome of patients with mCRC.

EGFR is expressed by most CRCs. Cetuximab (Erbitux) is a chimeric monoclonal antibody that specifically targets EGFR. In combination with Irinotecan, Cetuximab is approved for the treatment of EGFR-expressing mCRC, that has failed prior Irinotecan-based therapy, suggesting that Cetuximab may circumvent Irinotecan resistance.

Bevacizumab (Avastin) is a monoclonal antibody against Vascular Endothelial Growth Factor (VEGF). In CRC, increased VEGF expression correlates with invasiveness, vascular density, metastasis, recurrence and prognosis.

In a phase 2 trial of treatment of CRC, the addition of bevacizumab to FU/LV increased the response rate, the median time to disease progression, and the median duration of survival. Recently, it has been shown in randomized phase 2 trials that bevacizumab, when combined with irinotecan plus bolus FU/LV in the first line treatment of metastatic CRC, and with oxaliplatin plus continuous FU/LV (FOLFOX) in second-line treatment leads to an increased median survival, progression-free survival (PFS), and response rate compared with cytotoxic chemotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed locally advanced or metastatic colorectal cancer
* Measurable or evaluable disease according to the Response Evaluation Criteria in Solid Tumors (RECIST)
* ECOG performance status ≤ 2
* Age 18 - 72 years
* Patients who progress after 1st line therapy with FOLFOX/AVASTIN
* Adequate liver (Bilirubin ≤ 1.5 upper normal limit, SGOT/SGPT ≤ 4 upper normal limit, ALP ≤ 2.5 upper normal limit),renal (Creatinine ≤ 1.5 upper normal limit) and bone marrow (ANC ≥ 1,500/mm3, PLT ≥100,000/mm3) function
* Patients must be able to understand the nature of this study
* Written informed consent
* Previous treatments with all effective drugs for metastatic colorectal cancer (CPT-11, LOHP, 5-FU/XELODA, Erbitux, Avastin)

Exclusion Criteria:

* History of serious cardiac disease (unstable angina, congestive heart failure,uncontrolled cardiac arrhythmias)
* History of myocardial infarction or stroke within 6 months
* Clinically significant peripheral vascular disease
* History of abdominal fistula, gastrointestinal perforation or intraabdominal abscess within 28 days prior to Day 0
* Major surgical procedure, open biopsy, or significant traumatic injury within 30 days prior to Day 1
* Presence of central nervous system or brain metastases
* Evidence of bleeding diathesis or coagulopathy
* Blood pressure > 150/100 mmHg
* Pregnant or lactating woman
* Life expectancy < 3 months
* Previous radiotherapy within the last 4 weeks or > 25% of bone marrow
* Metastatic infiltration of the liver >50%
* Patients with chronic diarrhea (at least for 3 months) or partial bowel obstruction or total colectomy
* Active infection requiring antibiotics on Day 1
* Second primary malignancy, except for non-melanoma skin cancer and in situ cervical cancer
* Psychiatric illness or social situation that would preclude study compliance

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-10; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate | 3 - 6 month

SECONDARY OUTCOMES:
Time To Progression | 1 year
Toxicity profile | 28 days
Quality of life | 28 days
Symptoms improvement | 28 days
Overall Survival | Probability of 1-year survival (%)

CONTACTS AND LOCATIONS:
Overall Officials: Nikos Vardakis, MD, Principal Investigator — University Hospital of Crete, Dep of Medical Oncology
Locations (3):
- Greece (3):
  - University Hospital of Crete, Dep of Medical Oncology, Heraklion, Crete
  - University General Hospital of Alexandroupolis, Dep of Medical Oncology, Alexandroupoli
  - "IASO" General Hospital of Athens, 1st Dep of Medical Oncology, Athens